CLINICAL TRIAL: NCT00281294
Title: A Phase 2 Study to Evaluate the Safety, Tolerability, and Activity of Fontolizumab in Subjects With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early because the first phase didn't meet the endpoint.
Sponsor: PDL BioPharma, Inc. (Industry)
Organization: Facet Biotech (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZAF-711
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fontolizumab

INTERVENTIONS:
Drug: Fontolizumab

SUMMARY:
To evaluate the efficacy of fontolizumab in subjects with active rheumatoid arthritis as determined by a 50% improvement of an American College of Rheumatology criteria (ACR50) response at Week 14 (Stage A of study).

DETAILED DESCRIPTION:
To evaluate the efficacy of fontolizumab in subjects with active rheumatoid arthritis as determined by a 50% improvement of an American College of Rheumatology criteria (ACR50) response at Week 14 (Stage A of study).

Stage B of this trial is Double blind.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* A diagnosis of RA according to ACR criteria (Appendix D, American College of Rheumatology Clinical Classification Criteria for Rheumatoid Arthritis)
* RA functional class I, II, or III (Appendix E, ACR Revised Criteria for Classification of Functional Status in Rheumatoid Arthritis ) for at least 6 months
* Active RA with ≥ 6 tender joints and ≥ 6 swollen joints within one week of dosing or on Day 0, before dosing
* Serum CRP ≥ 1.0 mg/dL (10 mg/L) or ≥ 45 minutes of morning stiffness
* On stable doses for at least 30 days before receiving study drug of at least one, but not more than two, of the following disease-modifying antirheumatic drugs (DMARDs): hydroxychloroquine, leflunomide, methotrexate (leflunomide-methotrexate combination is unacceptable), or sulfasalazine. If being treated with nonsteroidal anti-inflammatory drugs (NSAIDs) or low-dose prednisone (≤ 10 mg/day), must be on stable regimen for at least 14 days before receiving study drug
* Women of childbearing potential with a negative serum pregnancy test at screening
* Subjects with reproductive potential agree to use a double-barrier method of contraception during the study and for 3 months after receiving last dose of study drug
* Must provide a signed and dated informed consent and an authorization to use protected health information, have the ability to understand the study requirements, and comply with study procedures, including required study visits

Exclusion Criteria:

* Significant involvement of secondary RA (eg, Felty's syndrome, pulmonary fibrosis, Sjogren's syndrome, vasculitis (keratoconjunctivitis sicca is not exclusionary)
* Received a live vaccine within 30 days of receiving fontolizumab
* Received an investigational agent within 30 days or five half-lives of the agent, whichever is longer, of receiving fontolizumab
* Received a corticosteroid injection into any joint, or has been treated with > 10 mg/day of a corticosteroid within 30 days of receiving fontolizumab
* Received etanercept or anakinra within 30 days of receiving fontolizumab
* Received gold salts, infliximab, or adalimumab within 60 days of receiving fontolizumab
* Received IV gamma-globulin or Prosorba column therapy within 90 days of receiving fontolizumab
* Received rituximab or cyclophosphamide within 6 months of receiving fontolizumab
* Failed B cell recovery after exposure to rituximab
* History of hypersensitivity to glycine, histidine, or Polysorbate 80
* Pregnant women or nursing mothers
* Malignancy within 5 years (excluding basal or squamous cell carcinoma of the skin or adequately treated cervical carcinoma in situ)
* Known chronic viral infections with HIV, hepatitis B, or hepatitis C
* Clinical, PPD, or clear radiographic evidence of prior TB
* Infection requiring hospitalization or parenteral medication, such as an antibiotic, antiviral, antifungal, or antiparasitic agent, within 90 days of receiving fontolizumab
* History of inflammatory joint disease (eg, gout, Lyme disease, psoriatic arthritis, reactive arthritis, seronegative spondyloarthropathy) or chronic inflammatory diseases (eg, inflammatory bowel disease, inflammatory myopathy, multiple sclerosis, overlap syndrome, scleroderma, systemic lupus erythematosus) other than RA
* Clinically significant unstable or poorly controlled acute or chronic diseases, such as myocardial infarction within 6 months, unstable angina, poorly controlled diabetes or hypertension
* ALT > 1.5 × the upper limit of normal; AST > 1.5 × the upper limit of normal; creatinine 1.5 × the upper limit of normal; absolute neutrophil count (ANC) < 1000/mm3; platelet count < 50,000/mm3
* History of any other medical disease, laboratory abnormalities, or psychological conditions that would make the subject (based upon the principal investigator's judgment) unsuitable for study enrollment
* Current abuse of alcohol or drugs (based upon investigator's assessment)
* Major surgery within 3 months prior to or planned elective surgery during or within 3 months after last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-12; Study Completion 2006-12

PRIMARY OUTCOMES:
-Proportion of subjects achieving an American College of Rheumatology response (ACR50) at Week 14 (Stage A).

SECONDARY OUTCOMES:
Proportion of subjects achieving ACR20, ACR50, and ACR70 (Stages A and B)
Change from baseline in serum CRP values (Stages A and B)
Percent improvement in individual ACR core outcome measures (Stages A and B)
Change from baseline in DAS28-CRP and ACR-N (Stages A and B)
ACR-N at each dosing day and at 1 and 3 months after the last dose of study drug (Stages A and B)
Number and proportion of subjects experiencing a disease flare-up since Week 14 (Stage B)
Time to disease flare since Week 14 (Stage B)
Assess the safety and tolerability of fontolizumab throughout the study by collection of the following:
Adverse events and SAEs up to 84 days after last dose of study drug; and, opportunistic or medically significant infections, malignancies, and onset of autoimmune diseases up to 6 months after last dose of study drug
Clinical laboratory measurements (hematology, serum chemistry) up to 84 days after last dose of study drug
Evaluation of pharmacokinetics (PK) up to 6 months after last dose of study drug (Stages A and B)
Evaluation of immunogenicity up to 6 months after last dose of study drug (Stages A and B)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C. Genovese, MD, Principal Investigator — Stanford University Medical Center-Div. of Rheumatology; Jerry Molitor, MD, PhD, Principal Investigator — Benaroya Research Institute at Virginia Mason; Michael H. Schiff, MD, Principal Investigator — Denver Arthritis Clinic; Alan Kivitz, MD, Principal Investigator — Altoona Center for Clinical Research; Craig Wiesenhutter, MD, Principal Investigator — Coeur d Alene Arthritis Clinic; Justus J. Fiechtner, MD, Principal Investigator — Justus Fiechtner MD PC; Daniel Wallace, MD, Principal Investigator — Wallace Rheumatic Study Center; Joel Kremer, MD, Principal Investigator — The Center for Rheumatology; Robert S. Katz, MD, Principal Investigator — Rheumatology Associates Clinical Research
Locations (9):
- United States (9):
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Stanford University Medical Center-Div. of Rheumatology, Palo Alto, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Coeur d Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Rheumatology Associates Clinical Research, Chicago, Illinois
  - Justus J. Fiechtner MD PC, Lansing, Michigan
  - The Center for Rheumatology, Albany, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington

REFERENCES:
- [Derived] Wilson JA, Prow NA, Schroder WA, Ellis JJ, Cumming HE, Gearing LJ, Poo YS, Taylor A, Hertzog PJ, Di Giallonardo F, Hueston L, Le Grand R, Tang B, Le TT, Gardner J, Mahalingam S, Roques P, Bird PI, Suhrbier A. RNA-Seq analysis of chikungunya virus infection and identification of granzyme A as a major promoter of arthritic inflammation. PLoS Pathog. 2017 Feb 16;13(2):e1006155. doi: 10.1371/journal.ppat.1006155. eCollection 2017 Feb. PMID 28207896